CLINICAL TRIAL: NCT02087358
Title: Alcohol Consumption and Stress at Patients Alcohol-dependants
Acronym: CASPA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P110908
Record Dates: First submitted 2014-02-24; First posted 2014-03-14 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Alcohol Dependence
Keywords: alcohol dependence; Stress- correlation; genetic; CRHR1
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CRHR1 gene polymorphisisme
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stress and craving: This 3 weeks study examines the correlation between stress and alcohol using an ecological, prospective design. Participants will be given phone calls 4 times a day for 3 weeks, assessing perceived stress and alcohol related craving.

SUMMARY:
This 3 weeks study examines the correlation between stress and alcohol using an ecological, prospective design.

DETAILED DESCRIPTION:
This 3 weeks study examines the correlation between stress and alcohol using an ecological, prospective design. Participants will be given phone calls 4 times a day for 3 weeks, assessing perceived stress and alcohol related craving.

ELIGIBILITY:
Inclusion criteria:

* Males or Females aged 18-65 years
* Alcohol use disorder defined by DSM 5 criteria
* Fluent in French
* Hospitalized for alcohol withdrawal for at least 7 days
* Viable (working) telephone number

Exclusion criteria:

* Participants without social care insurance
* Any DSM Axis I disorder not defined in the inclusion criteria
* Mandatory psychiatric treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes alcohol dependent inpatients participating in a 3 weeks detoxification program.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-07; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Stress level | 3 weeks follow-up
  correlation between stress and alcohol related craving using a prospective ecological design

SECONDARY OUTCOMES:
Genetic association with stress level | 3 weeks follow-up
  Correlation between stress and alcohol related craving using a prospective ecological design stratified for CRHR1 variant

CONTACTS AND LOCATIONS:
Overall Officials: Yann Le Strat, Pr MD, Principal Investigator — Psychiatrist Service
Locations (1):
- Hopital Louis Mourier, Service de psychiatrie, Colombes, France